CLINICAL TRIAL: NCT06250166
Title: Feasibility, Acceptability, and Effectiveness of an Individualized Plant-based (iPLANT) Diet Plan in Colorectal Cancer: Mixed Method Embedded Design
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Malaysia (Other Government)
Responsible Party: Principal Investigator, Krystal Ng Lu Shin, Principal Investigator, National Cancer Institute, Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-00024-WJG
Record Dates: First submitted 2024-02-01; First posted 2024-02-08 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer; Nutrition Poor; Gastrointestinal Complication; Quality of Life
MeSH Terms: conditions — Colorectal Neoplasms; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Receive iPLANT diet plan and diet counselling by a qualified dietitian in oncology setting.
  Interventions: Behavioral: iPLANT diet plan and diet counselling
- Control group (Active Comparator): Receive usual diet counselling only
  Interventions: Behavioral: Usual diet counselling

INTERVENTIONS:
Behavioral: iPLANT diet plan and diet counselling — A diet plan which mainly consists of plant-based food will be designed based on participants' energy and protein needs. The counselling covers (1) guidance to achieve energy and protein requirement (2) advice on food to be included in iPLANT diet plan (Mediterranean diet: increase intake of fish and legumes; moderate intake of eggs, dairy, nuts, poultry; limit intake of red meat).
  Arms: Intervention group
Behavioral: Usual diet counselling — General dietary advices on how to improve oral intake and maintain healthy weight will be provided.
  Arms: Control group

SUMMARY:
The goal of this intervention study is to investigate the effectiveness of individualized plant-based diet plan on nutritional indices and clinical outcomes in colorectal cancer patients receiving chemotherapy. The main questions to answer are:

1. What are the current eating trends in colorectal cancer patients?
2. What are the common perceptions of adopting a plant-based diet in colorectal cancer?
3. Does iPLANT diet plan improve nutritional indices of colorectal cancer patients?
4. Does iPLANT diet plan improve patients' gastrointestinal side effects and quality of life without compromising their nutritional status?

Participants will be randomly assigned into two arms (intervention and control) using opaque envelop system. Intervention group will receive individualized plant-based diet plan and diet counselling, whereas the control group will receive usual diet counselling.

The researcher will compare the differences in nutritional outcomes and quality of life between intervention and control groups before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with colorectal cancer, including the sites of caecum, appendix, ascending colon, hepatic flexure, transverse colon, splenic flexure, descending colon, sigmoid colon, and rectum
* TNM stage II to IV
* Receiving chemotherapy
* Able to take food orally

Exclusion Criteria:

* Have cognitive impairments or mental disorders
* Diagnosed with severe illness, such as chronic kidney disease and chronic obstructive pulmonary disease
* Within 4 weeks of bowel resection
* Terminally ill or receive hospice care
* Receiving enteral or total parenteral nutrition
* Having inflammatory bowel diseases
* Having gastrointestinal bleeding or obstruction
* Pregnancy or breastfeeding
* Severe anemia (<0.8g/dL)
* ECOG performance score >2
* High stoma output (>1500ml per day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mean Prognostic Nutritional Index at 12 weeks | Change from baseline to week 12
  The Prognostic Nutritional Index is used to assess the nutritional status. Respondents are severely malnourished if score less than 40
Change from baseline in mean neutrophil-lymphocyte ratio at 12 weeks | Change from baseline to week 12
  Higher score indicates higher level of inflammation
Change from baseline in mean platelet-lymphocyte ratio at 12 weeks | Change from baseline to week 12
  Higher score indicates higher level of inflammation

SECONDARY OUTCOMES:
Change from baseline in mean Patient-Generated Subjective Global Assessment score at 12 weeks | Change from baseline to week 12
  The PG-SGA score is derived from components of weight history, food intake, nutritional impact symptoms, and activity function. The possible scores range from 0 (well-nourished) to 37 (worst possible malnourished)
Change from baseline in mean skeletal muscle Index, body fat mass, extracellular water ratio, phase angle at 12 weeks | Change from baseline to week 12
  The higher values of skeletal muscle index and phase angle indicate lower risk of malnutrition, whereas higher reading of extracellular water ratio indicates higher risk of malnutrition. Higher body fat mass indicates higher adiposity level.
Change from baseline in mean mid arm muscle area at 12 weeks | Change from baseline to week 12
  Respondents develop cachexia if values are less than 32 (male) and 18 (female)
Change from baseline in mean handgrip strength at 12 weeks | Change from baseline to week 12
  Respondents have weak muscle if the values are 27 or less (male) and 16 or less (female)
Change from baseline in mean quality of Life at 12 weeks | Change from baseline to week 12
  EORTC QLQ-CR29 is a validated tool to measure the functional scales and symptomatic level of colorectal cancer that resulted from disease or treatment factors. Possible scores range from 0 to 100, which higher score indicates better functional scale or worse symptomatic level
Change in mean daily energy and protein intake at 12 weeks | Change from baseline to week 12
  Higher intake of daily energy and protein indicates improved oral intake

CONTACTS AND LOCATIONS:
Locations (2):
- Malaysia (2):
  - Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - National Cancer Institute, Putrajaya, Putrajaya

IPD SHARING:
Plan to Share IPD: No